CLINICAL TRIAL: NCT04664244
Title: Combination of Nimotuzumab and Radiotherapy for Recurrent and Metastatic Uterine Cervical Squamous Carcinoma: a Single-arm, Open, Phase 2 Clinical Trial
Brief Title: Combination of Nimotuzumab and Radiotherapy for Recurrent Uterine Cervical Squamous Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lei Li (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-NIMO1
Record Dates: First submitted 2020-12-05; First posted 2020-12-11 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Recurrent Cervical Carcinoma; Radiotherapy; Epidermal Growth Factor Receptor; Nimotuzumab; Objective Response Rate; Progression-free Survival; Overall Survival
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Intervention Model Description: All eligible patients will undergo the same treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All eligible patients (Experimental): All eligible patients enrolled
  Interventions: Combination Product: Combination of nimotuzumab and radiotherapy

INTERVENTIONS:
Combination Product: Combination of nimotuzumab and radiotherapy — Patients will undergo targeted radiotherapy no more than 8 weeks, and concurrent nimotuzumab 200 mg intravenous injection every one week till the ending of radiotherapy. Then patients undergo a maintaining therapy with nimotuzumab 200 mg intravenous injection every two weeks up to one year or till the disease progresses.

SUMMARY:
Patients with recurrent or metastatic uterine cervical squamous carcinoma have very poor prognosis. For eligible patients, radiotherapy remains the choice, which has the most effective impact on the survival periods. On the hand, anti-angiogenic therapy has been proved to be promising treatment for recurrent or advanced cervical carcinomas. This study aims to discover the objective response of combination therapy with nimotuzumab (an anti-epidermal growth factor receptor [EGFR] IgG1 humanized monoclonal antibody) and radiotherapy in recurrent or metastatic uterine cervical squamous carcinoma in a single-arm, open, phase 2 clinical trial. The primary endpoint is the objective response rate evaluated by imaging methods. The second endpoints are the progression-free survival and overall survival. The treatment toxicity is regarded as one the second endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Female aged more than 18 years
* Eastern Cooperative Oncology Group score 0-1
* Pathological confirmed of uterine cervical squamous carcinoma
* An interval of 3 months or more since the fulfilling of last treatment
* At least one measurable lesion defined by Response Evaluation Criteria in Solid Tumors (RECIST) guideline 1.1
* Anticipative survival period of 3 months or more
* Lab testing within reference ranges
* With appropriate contraception
* Provided consents of participating the trial

Exclusion Criteria:

* With a history of exposure to other antiangiogenic agents
* With other malignancies within past 3 years
* With vital complications
* With uncontrolled hypertension despite of medical treatment
* With brain metastasis
* With addiction to psychiatric medications or with mental disorders

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2020-12-19 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 1 years
  The objective response rate includes complete and partial remission

SECONDARY OUTCOMES:
Progression-free survival | 2 years
  Progression-free survival from the end of radiotherapy to the disease progression
Overall survival | 3 years
  Overall survival from the start of radiotherapy to the disease progression
Disease control rate | 1 year
  The rates of complete and partial remission, and stable disease
Adverse event rates | 3 years
  The rates of adverse events judged by Common Terminology Criteria for Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Lei Li, Beijing, Beijing Municipality, China